CLINICAL TRIAL: NCT07124949
Title: Chinese Migrant Population Health Cohort
Status: Recruiting | Type: Observational
Sponsor: Jinwei Tian (Other)
Collaborators: Hainan Medical College (Other)
Responsible Party: Sponsor-Investigator, Jinwei Tian, Doctor, Harbin Medical University
Organization: Harbin Medical University (Other)
Other Study IDs: HMUIRB2024029PRE; ZY04JD01 (Other Grant/Funding Number: The Project of the Central Governmen Funds for Guiding Local Science and Technology Development in Heilongjiang Provinc)
Record Dates: First submitted 2025-08-11; First posted 2025-08-15 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases; Metabolic Disorders; Ageing and Geriatric Health; Climate Adaptation
Keywords: Cardiovascular Diseases; Metabolic Diseases; Geriatrics; Migration; Climate Change; Health Promotion
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood (serum, plasma, buffy coat, and peripheral blood mononuclear cells), urine, stool, hair, and nail samples will be collected and stored. Blood samples will be processed for biochemical assays, DNA, RNA, and multi-omics analyses (including metabolomics, proteomics, and lipidomics). Urine and stool samples will be analyzed for metabolic, microbiome, and environmental exposure markers. Hair and nail samples will be used for long-term exposure assessment (e.g., heavy metals, stable isotopes). All biospecimens will be stored in a certified biobank at -80 °C for future research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Winter Migrant Group: No Intervention
  Interventions: Other: No intervention
- Summer Migrant Group: No Intervention
  Interventions: Other: No intervention
- Cold-Region Resident Group: no Intervention
  Interventions: Other: No intervention
- Tropical-Region Resident Group: no Intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — no intervention

SUMMARY:
The Chinese Migrant Population Health Cohort is a prospective, multi-center study jointly initiated by Professor Yong Ji, President of Harbin Medical University, and Academician Guoqiang Chen, President of Hainan Medical University, in collaboration with regional partners. It targets older adults (≥60 years) who engage in seasonal migration between cold (Heilongjiang) and tropical (Hainan) regions. The primary objective is to investigate cardiovascular and metabolic disease risks, underlying biological and environmental mechanisms, and effective preventive strategies in this unique population.

Participants are recruited from both origin and destination sites and undergo standardized baseline assessments, including questionnaires, physical examinations, medical imaging, biospecimen collection (blood, stool, hair, nails), and environmental exposure monitoring. Longitudinal follow-up includes periodic reassessments, remote monitoring, and data linkage with hospital information systems to capture health outcomes.

The study aims to:

Define migration-related health risk profiles and disease phenotypes.

Elucidate biological and environmental mechanisms influencing disease onset and progression.

Develop AI-driven risk prediction models and evaluate targeted interventions through nested randomized controlled trials.

Translate findings into clinical guidelines and scalable cross-regional health management models.

This is the first cohort in China to systematically investigate the health impacts of seasonal migration in older adults. By integrating epidemiology, multi-omics, environmental data, and health policy translation, the study seeks to improve continuity of care, strengthen climate adaptation, and promote healthy ageing.

ELIGIBILITY:
Inclusion Criteria:

1. Permanent residents of Harbin or Hainan who will continue to reside in Harbin or Hainan for the next 5 years.
2. Baseline age ≥60 years, with basic communication and comprehension abilities.
3. No confirmed diagnosis of end-stage major organic diseases (e.g., advanced heart failure, advanced liver failure, advanced kidney failure, malignant tumors).
4. Able to perform activities of daily living independently and capable of completing questionnaires and physical examinations.
5. Willing to participate in the study, provide written informed consent, accept long-term follow-up, and provide biological specimens.

Exclusion Criteria:

1. Occurrence of life-threatening acute events (e.g., myocardial infarction, acute heart failure, stroke) within the past 30 days.
2. Currently receiving chronic treatment with antiviral drugs (e.g., for HIV) or antipsychotic medications.
3. Presence of moderate to severe cognitive impairment preventing survey completion or follow-up cooperation.
4. Current acute infectious diseases such as influenza or fever.
5. Simultaneous participation in other interventional clinical studies.
6. Refusal to sign informed consent or unwillingness to provide biological specimens.
7. Any other condition deemed unsuitable for study participation by the investigators based on overall assessment.

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will enroll community-dwelling adults aged ≥60 years from Harbin (cold region) and Hainan (tropical region), China. Four groups will be included: 1. Winter Migrant Group: ~5,000 Harbin residents who habitually migrate to Hainan during the cold season for ≥2 months each time, with ≥2 consecutive years of such migration and plans to continue; 2. Summer Migrant Group: ~1,000 Hainan residents who habitually migrate to Harbin during the hot season for ≥2 months, with similar migration history and plans; 3. Cold-Region Resident Group: ~10,000 Harbin residents, including matched controls for migrant groups and randomly selected residents, with no >2 months residence outside Harbin in the past 5 years; 4. Tropical-Region Resident Group: ~10,000 Hainan residents with similar matching criteria and residency requirements.
  All participants must be able to communicate, perform daily activities independently, consent to long-term follow-up, and provide biospecimens.
Sampling Method: Non-Probability Sample
Enrollment: 26000 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing First Major Cardiovascular Event | Up to 5 years from baseline
  First occurrence of myocardial infarction, stroke (ischemic or hemorrhagic), or cardiovascular death, confirmed through hospital records, death registries, and adjudication committee review.

SECONDARY OUTCOMES:
Number of Participants with New-Onset Metabolic Disorders | Up to 5 years from baseline
  New-onset type 2 diabetes mellitus, dyslipidemia, or obesity as defined by standard clinical and laboratory criteria.
Number of Deaths from Any Cause | Up to 5 years from baseline
  Death from any cause, verified through official death certificates and hospital records.
Changes in Cardiometabolic Risk Factors | Baseline, 2 years, 4 years
  Longitudinal changes in blood pressure, fasting glucose, HbA1c, lipid profile, BMI, waist circumference, and body composition.
Change in EQ-5D Quality of Life Score from Baseline | Baseline, 2 years, 4 years
  Changes in validated quality-of-life scales (e.g., EQ-5D).
Change in Cognitive Function Score (MoCA) from Baseline | Baseline, 2 years, 4 years
  Mean change in Montreal Cognitive Assessment score.

OTHER OUTCOMES:
Change in Carotid Intima-Media Thickness from Baseline | Baseline and follow-up imaging
  Mean change (mm) measured by carotid ultrasound.
Change in Coronary Artery Calcium Score from Baseline | Baseline and follow-up imaging
  Mean change in Agatston score by CT angiography.
Change in Plasma Metabolite Levels from Baseline | Baseline and follow-up biospecimen analyses
  Relative or absolute change in concentrations of targeted metabolites identified through mass spectrometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oswald R. NHS ombudsman. A job for strife. Health Serv J. 1998 Oct 8;108(5625):30-1. PMID 10186180
- [Background] Ebert MP, Hoffmann J, Haeckel C, Rutkowski K, Schmid RM, Wagner M, Adler G, Schulz HU, Roessner A, Hoffmann W, Malfertheiner P. Induction of TFF1 gene expression in pancreas overexpressing transforming growth factor alpha. Gut. 1999 Jul;45(1):105-11. doi: 10.1136/gut.45.1.105. PMID 10369712
- [Background] Sesso Rde C, Ajzen H. [Treatment with dialysis of chronic renal patients]. Rev Assoc Med Bras (1992). 1995 Jan-Feb;41(1):1-2. No abstract available. Portuguese. PMID 7550406
- [Background] Compliance interventions make a difference, but focus should shift to patient outcomes. Am J Health Syst Pharm. 1998 Nov 1;55(21):2231. doi: 10.1093/ajhp/55.21.2231. No abstract available. PMID 9825873
- [Background] Sasieni P. Cervical screening: what is the point? Lancet. 1995 Jul 22;346(8969):244; author reply 246-7. No abstract available. PMID 7616810
- [Background] Kobayashi T, Kimura T, Yoshida M, Sakuramachi S, Takeuchi Y, Harada Y, Suzuki K, Ishikawa A. [A case of rectal cancer in adenoma diagnosed 7 years after renal transplantation]. Nihon Shokakibyo Gakkai Zasshi. 1996 Oct;93(10):738-42. No abstract available. Japanese. PMID 8921708
- [Background] Focht S. Spirituality becomes a prominent component of holistic care. Oncol Nurs Forum. 1998 Jul;25(6):988-90. No abstract available. PMID 9679254
- [Background] Kudla G, Montessuit S, Eskes R, Berrier C, Martinou JC, Ghazi A, Antonsson B. The destabilization of lipid membranes induced by the C-terminal fragment of caspase 8-cleaved bid is inhibited by the N-terminal fragment. J Biol Chem. 2000 Jul 28;275(30):22713-8. doi: 10.1074/jbc.M003807200. PMID 10801880
- [Background] Hanada K, Song CZ, Yamamoto K, Yano K, Maeda Y, Yamaguchi K, Muramatsu M. RNA polymerase I associated factor 53 binds to the nucleolar transcription factor UBF and functions in specific rDNA transcription. EMBO J. 1996 May 1;15(9):2217-26. PMID 8641287
- [Background] Tsunemi K, Nishimoto M, Takai S, Yuda A, Nishimoto Y, Hasegawa S, Asada K, Sawada Y, Kondo K, Fukumoto H, Miyazaki M, Sasaki S. [Role of angiotensin II-forming pathway in ruptured aortic aneurysms]. Nihon Geka Gakkai Zasshi. 2001 Feb;102(2):243. No abstract available. Japanese. PMID 11260908
- [Background] Piperberg JB, Reif-Lehrer L. Glutamine synthetase in cultured whole retinas from the embryonic chick. Role of protein and RNA syntheses in 4 degrees C storage enhancement. Cell Biophys. 1984 Jun;6(2):131-48. doi: 10.1007/BF02788592. PMID 6207921
- [Background] Finnish Gastroenterological Association's work group. [Endoscopic retrograde cholangiopancreatography]. Duodecim. 1999;115(11):1262-7. No abstract available. Finnish. PMID 11877845
- [Background] Canziani R, Bertoni PD, Arancio F, Boghi M, Zanetti A, Binaghi G. [Evaluation of coronary risk factors in a 30-year-old population from the province of Varese]. Cardiologia. 1982;27(7):697-705. No abstract available. Italian. PMID 6927500
- [Background] Berglund B. High-altitude training. Aspects of haematological adaptation. Sports Med. 1992 Nov;14(5):289-303. doi: 10.2165/00007256-199214050-00002. PMID 1439397
- [Background] Fernandez S, Arce G, Garcia-Alaminos A, Cazcarro I, Arto I. Climate change as a veiled driver of migration in Bangladesh and Ghana. Sci Total Environ. 2024 Apr 20;922:171210. doi: 10.1016/j.scitotenv.2024.171210. Epub 2024 Feb 26. PMID 38417512
- [Background] Cao B, Bai C, Wu K, La T, Su Y, Che L, Zhang M, Lu Y, Gao P, Yang J, Xue Y, Li G. Tracing the future of epidemics: Coincident niche distribution of host animals and disease incidence revealed climate-correlated risk shifts of main zoonotic diseases in China. Glob Chang Biol. 2023 Jul;29(13):3723-3746. doi: 10.1111/gcb.16708. Epub 2023 Apr 17. PMID 37026556
- [Background] Briggs S, Cavet J, Lamb C, Lightowlers S. Cancer and climate change: the environmental impact of cancer care. Lancet Oncol. 2021 Feb;22(2):e38. doi: 10.1016/S1470-2045(20)30740-3. No abstract available. PMID 33539745
- [Background] Vicedo-Cabrera AM, Melen E, Forastiere F, Gehring U, Katsouyanni K, Yorgancioglu A, Ulrik CS, Hansen K, Powell P, Ward B, Hoffmann B, Andersen ZJ. Climate change and respiratory health: a European Respiratory Society position statement. Eur Respir J. 2023 Sep 3;62(2):2201960. doi: 10.1183/13993003.01960-2022. Print 2023 Aug. No abstract available. PMID 37661094
- [Background] Jiang Y, Hu J, Peng L, Li H, Ji JS, Fang W, Yan H, Chen J, Wang W, Xiang D, Su X, Yu B, Wang Y, Xu Y, Wang L, Li C, Chen Y, Zhao D, Kan H, Ge J, Huo Y, Chen R. Non-optimum temperature increases risk and burden of acute myocardial infarction onset: A nationwide case-crossover study at hourly level in 324 Chinese cities. EClinicalMedicine. 2022 Jun 17;50:101501. doi: 10.1016/j.eclinm.2022.101501. eCollection 2022 Aug. PMID 35755601
- [Background] Khraishah H, Alahmad B, Ostergard RL Jr, AlAshqar A, Albaghdadi M, Vellanki N, Chowdhury MM, Al-Kindi SG, Zanobetti A, Gasparrini A, Rajagopalan S. Climate change and cardiovascular disease: implications for global health. Nat Rev Cardiol. 2022 Dec;19(12):798-812. doi: 10.1038/s41569-022-00720-x. Epub 2022 Jun 7. PMID 35672485
- [Background] Zhang S, Zhang C, Cai W, Bai Y, Callaghan M, Chang N, Chen B, Chen H, Cheng L, Dai H, Dai X, Fan W, Fang X, Gao T, Geng Y, Guan D, Hu Y, Hua J, Huang C, Huang H, Huang J, Huang X, Ji JS, Jiang Q, Jiang X, Kiesewetter G, Li T, Liang L, Lin B, Lin H, Liu H, Liu Q, Liu X, Liu Z, Liu Z, Liu Y, Lu B, Lu C, Luo Z, Ma W, Mi Z, Ren C, Romanello M, Shen J, Su J, Sun Y, Sun X, Tang X, Walawender M, Wang C, Wang Q, Wang R, Warnecke L, Wei W, Wen S, Xie Y, Xiong H, Xu B, Yan Y, Yang X, Yao F, Yu L, Yuan J, Zeng Y, Zhang J, Zhang L, Zhang R, Zhang S, Zhang S, Zhao M, Zheng D, Zhou H, Zhou J, Zhou Z, Luo Y, Gong P. The 2023 China report of the Lancet Countdown on health and climate change: taking stock for a thriving future. Lancet Public Health. 2023 Dec;8(12):e978-e995. doi: 10.1016/S2468-2667(23)00245-1. Epub 2023 Nov 18. No abstract available. PMID 37989307